CLINICAL TRIAL: NCT03768856
Title: Feasibility Study of Temporally Feathered Radiation Therapy (TFRT) for Head and Neck Squamous Cell Carcinoma: Means of Toxicity Reduction
Brief Title: Temporally Feathered Radiation Therapy (TFRT) for Head and Neck Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE4318
Record Dates: First submitted 2018-11-13; First posted 2018-12-07 (Actual); Results first posted 2020-07-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Head and Neck Cancer
Keywords: Radiation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Temporally Feathered Radiation Therapy (TFRT) (Experimental): Temporally feathered radiation therapy is designed for targets within close proximity to multiple organs at risk. The foundation of this planning technique is the rotation of radiation dose to the nearby organs at risk on a daily basis, and hence the term "feathering".
  Interventions: Radiation: Temporally Feathered Radiation Therapy (TFRT)

INTERVENTIONS:
Radiation: Temporally Feathered Radiation Therapy (TFRT) — Up to 5 different plans are created and delivered on a daily basis Monday-Friday for 7 weeks. The treating physician designates up to 5 organs at risk (OARs) to be feathered based on the proximity to the target. The daily prescription dose delivered to the Planning Target Volumes (PTV) is not changed.

SUMMARY:
This study will evaluate the feasibility of using more advanced IMRT (intensity modulated radiation therapy) techniques. This new technique is termed Temporally Feathered Radiation Therapy (TFRT). TFRT is designed to reduce the side effects of conventional radiation therapy. Research has shown that TFRT may lessen these side effects.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the feasibility of TFRT planning and delivery for head and neck squamous cell carcinoma. Secondary objectives include estimating grade 3-5 acute toxicity (within 90 days) and describing patient-reported outcomes (PRO) of toxicity during and after TFRT. This study is planned as a single arm feasibility trial to demonstrate clinical delivery of TFRT plans. Five patients will be accrued as a single cohort.

When using standard-of-care intensity modulated radiation therapy (IMRT), a single radiation plan is created and delivered on a daily basis Monday-Friday for a total of 7 weeks. In contrast, when using TFRT, up to 5 different plans are created and delivered each specific day of the week. Treatments will still occur on a daily basis Monday-Friday for 7 weeks. In each of these radiation plans used for TFRT, the radiation dose that will be delivered to the nearby healthy tissues will vary, allowing for increased time for normal tissue to recover from radiation-induced damage. Once weekly, a slightly higher radiation dose will be delivered to the "feathered" organ. On the remaining four days of the week, a slightly lower radiation dose will be delivered to the "feathered" organ. The radiation dose that will be delivered to the areas of cancer will not be changed. In this study, only the radiation dose delivered to the normal healthy tissues will be changed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically or cytologically confirmed squamous cell carcinoma arising from a primary head and neck site (oral cavity, oropharynx, larynx/hypopharynx, nasopharynx).TX-4, NX-3, MX-0 stages are permitted.
* Subjects must be eligible for definitive radiation therapy (70Gy in 35 fractions) with or without chemotherapy.
* Karnofsky Performance status ≥80.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Subjects receiving any other investigational agents.
* Postoperative radiotherapy is not permitted.
* History of prior head and neck radiation therapy.
* Subjects with uncontrolled inter-current illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or breastfeeding women are excluded from this study because radiation therapy has the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with radiation therapy, breastfeeding should be discontinued if the mother is treated with radiation therapy. These potential risks may also apply to other agents used in this study.
* The patient cannot have distant metastatic disease (or M1 disease by AJCC 8th edition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-12-07 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nikhil Joshi, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants enrolled in study
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 5
Age, Customized [Count of Participants; unit: Participants]
  50-59 years | 2
  60-69 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of TFRT Planning and Delivery Defined by Number of Participants Starting Radiotherapy Within 15 Days of Simulation
Description: Number of participants starting radiotherapy within 15 days of simulation. The TFRT technique will be deemed feasible if 3/5 participants meet this criteria.
Time Frame: 15 days from start of treatment
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 5
Participants | 4

2. Secondary Outcome: Number of Participants Who Experienced Grade 3-5 Acute Toxicities Per CTCAE Version 4
Description: Number of participants who experienced grade 3-5 acute toxicities as defined by CTCAE version 4
Time Frame: Up to 90 days after treatment
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 5
Participants | 1

3. Secondary Outcome: Participant-reported Outcomes (PRO) During TFRT Using EORTC QLQ-C30 Questionnaire
Description: Global health status/health-related quality of life measurements based on European Organization of Research and Treatment Of Cancer tool general (EORTC QLQ-H&N35). Scores range from 0-100.
Time Frame: At weeks 1, 4, and 7 of treatment and at 2 weeks, 4 weeks, and 3 months post-treatment
Population: No participant were analyzed for quality of life questionnaires as there was an error in obtaining this data. A trial deviation was filed for this error.
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 0

4. Secondary Outcome: Participant-reported Outcomes (PRO) During TFRT Using EORTC QLQ-H&N35 Questionnaire
Description: Health-related quality of life measurements and symptoms among head and neck cancer participants based on European Organization of Research and Treatment of Head and Neck cancer questionnaire (EORTC QLQ-C30). Scores range from 0-100.
Time Frame: At weeks 1, 4, and 7 of treatment and at 2 weeks, 4 weeks, and 3 months post-treatment
Population: No participants were analyzed for quality of life questionnaires as there was an error in obtaining this data. A trial deviation was filed for this error.
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 0

5. Secondary Outcome: Participant-reported Outcomes (PRO) of Mouth Dryness After TFRT Using Xerostomia Questionnaire
Description: Xerostomia Questionnaire is a questionnaire used to describe mouth dryness and its effects on daily life. Scores range from 0-100. A high score represents a worse Xerostomia.
Time Frame: At week 1, 4, and 7 of treatment and at 2 weeks, 4 weeks, and 3 months post-treatment
Population: as for outcome 4
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants Considered Compliant With Plan Delivery
Description: Number of participants who were able to complete the treatment course within the allotted time and without deviations and complete the questionnaires within the allotted time. Considered successful if 3/5 complete prescribed treatment course per protocol.
Time Frame: 5 months from start of treatment
Population: Participants enrolled in study
Measure: Count of Participants; unit: Participants
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
Number analyzed (Participants) | 5
Participants | 4

ADVERSE EVENTS:
Time Frame: Up to 3 mos post post-treatment
Arm/Group | Temporally Feathered Radiation Therapy (TFRT)
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temporally Feathered Radiation Therapy (TFRT) (N=5)
Acute kidney injury (Endocrine disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-08): https://cdn.clinicaltrials.gov/large-docs/56/NCT03768856/Prot_SAP_002.pdf
  • Informed Consent Form (2019-10-26): https://cdn.clinicaltrials.gov/large-docs/56/NCT03768856/ICF_001.pdf